CLINICAL TRIAL: NCT02447809
Title: The Association Between Plasma or Platelet microRNAs and Clopidogrel Low Response and Its Mechanism
Brief Title: Plasma and Platelet microRNAs in Clopidogrel Low Response Patients
Acronym: PPRC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Chunjian Li, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 004
Record Dates: First submitted 2015-05-05; First posted 2015-05-19 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Coronary Artery Disease
Keywords: microRNA; Platelet; Clopidogrel low response
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regular DAPT(IPA≤60%) (Experimental): ASA and Clopidogrel
  Interventions: Drug: Clopidogrel; Drug: acetylsalicylic acid (ASA)
- Regular DAPT(IPA>60%) (Active Comparator): ASA and Clopidogrel
  Interventions: Drug: Clopidogrel; Drug: acetylsalicylic acid (ASA)

INTERVENTIONS:
Drug: Clopidogrel — (ASA 100mg daily and Clopidogre 75mg daily)* 12 month.
  Other Names: Plavix
Drug: acetylsalicylic acid (ASA)

SUMMARY:
Clopidogrel is an important anti-platelet agent.However, about 30% of the coronary artery disease patients presented clopidogrel low response (CLR).Previous studies showed that the cardiovascular event ratio of the CLR patients was 4.4 times of the normal responders.

It is known that the plasma and platelet miRNAs are determined by different disease status when platelets are released from the megakaryocyte, and the platelet miRNAs can adjust the expressions of the platelet's receptors and proteins.The purpose of this study is to find multiple platelet miRNAs involved in the development of CLR, and platelet miRNAs cause CLR through adjusting the expressions of the key receptors and proteins in the ADP activating pathway and consequently reducing their responses to clopidogrel.

The CLR will be detected by light transmission aggregometry (LTA) and vasodilator-stimulated phosphoprotein phosphorylation (VASP-P). Differential expressions of plasma and platelet miRNAs profile in CLR patients will be screened by deep sequencing and validated to investigate the association between plasma and platelet miRNAs profile and CLR as well as the patients' prognosis.The study results would serve as markers for individualized anti-platelet treatment, and supply new targets for the treatment of coronary artery disease.

DETAILED DESCRIPTION:
A multiphase, case-control study was designed to identify plasma and platelet miRNAs as surrogate markers for CLR .

All patients take 300mg loading dose clopidogrel plus 100mg daily ASA and 75mg daily clopidogrel after admission. Patients are recruited after percutaneous coronary intervention (PCI). Light transmittancy aggregation (LTA) in response to 5μM ADP is to measured 5 days after taking the loading dose clopidogrel.Than CLR patients were selected.

In the initial biomarker-screening stage, plasma and platelet samples from 20 CLR patients and 20 controls underwent Solexa sequencing to identify miRNAs that showed significant differences between the CLR cases and matched controls.

Subsequently,we performed a biomarker confirmation analysis with a hydrolysis probe-based RT-qPCR assay to refine the number of plasma and platelet miRNAs in the CLR signature. This analysis was carried out in 2 phases: (a) the biomarker-selection phase, in which plasma and platelet samples from 20 CLR patients and 20 control individuals formed the training set, and (b) the biomarker-validation phase, in which plasma and platelet samples from an additional 80 CLR patients and 80 controls formed the validation set.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive stent implantation;
* Patients who take 100mg daily ASA and 75mg daily clopidogrel
* Patient age >18 years and <80 years old;
* Signed inform consent

Exclusion Criteria:

* Allergy or intolerance to ASA,clopidogrel;
* Patients who are planning to take warfarin or drugs that potentially could interfere with the anti-platelet effects of ASA,clopidogrel.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The expressions of miRNAs profile | 5-days After recruited
  Two pools of plasma and platelet were collected from participants separately. The total RNA of each pool was extracted by using Trizol Reagent. An initial screening of miRNAs expression was performed by Solexa sequencing. And differential expression was validated using RT-qPCR in individuals samples.

SECONDARY OUTCOMES:
Clinical efficacy | 1-month and 1-year after recruited
  1-month and 1-year death,non-fatal myocardial infarction,ischemic stroke,revascularization and stent thrombosis(ARC definition)

OTHER OUTCOMES:
Bleeding | 1-month and 1-year after recruited
  1-month and 1-year minor,moderate and major bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Chunjian Li, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Yusuf S, Zhao F, Mehta SR, Chrolavicius S, Tognoni G, Fox KK; Clopidogrel in Unstable Angina to Prevent Recurrent Events Trial Investigators. Effects of clopidogrel in addition to aspirin in patients with acute coronary syndromes without ST-segment elevation. N Engl J Med. 2001 Aug 16;345(7):494-502. doi: 10.1056/NEJMoa010746. PMID 11519503
- [Background] Siller-Matula JM, Trenk D, Schror K, Gawaz M, Kristensen SD, Storey RF, Huber K; EPA (European Platelet Academy). Response variability to P2Y12 receptor inhibitors: expectations and reality. JACC Cardiovasc Interv. 2013 Nov;6(11):1111-28. doi: 10.1016/j.jcin.2013.06.011. PMID 24262612
- [Background] Calin GA, Croce CM. MicroRNA-cancer connection: the beginning of a new tale. Cancer Res. 2006 Aug 1;66(15):7390-4. doi: 10.1158/0008-5472.CAN-06-0800. PMID 16885332
- [Background] Hu Z, Chen X, Zhao Y, Tian T, Jin G, Shu Y, Chen Y, Xu L, Zen K, Zhang C, Shen H. Serum microRNA signatures identified in a genome-wide serum microRNA expression profiling predict survival of non-small-cell lung cancer. J Clin Oncol. 2010 Apr 1;28(10):1721-6. doi: 10.1200/JCO.2009.24.9342. Epub 2010 Mar 1. PMID 20194856
- [Background] Clancy L, Freedman JE. New paradigms in thrombosis: novel mediators and biomarkers platelet RNA transfer. J Thromb Thrombolysis. 2014 Jan;37(1):12-6. doi: 10.1007/s11239-013-1001-1. PMID 24163053
- [Background] Landry P, Plante I, Ouellet DL, Perron MP, Rousseau G, Provost P. Existence of a microRNA pathway in anucleate platelets. Nat Struct Mol Biol. 2009 Sep;16(9):961-6. doi: 10.1038/nsmb.1651. Epub 2009 Aug 9. PMID 19668211
- [Background] Dangelmaier C, Jin J, Smith JB, Kunapuli SP. Potentiation of thromboxane A2-induced platelet secretion by Gi signaling through the phosphoinositide-3 kinase pathway. Thromb Haemost. 2001 Feb;85(2):341-8. PMID 11246558
- [Background] Li C, Fang Z, Jiang T, Zhang Q, Liu C, Zhang C, Xiang Y. Serum microRNAs profile from genome-wide serves as a fingerprint for diagnosis of acute myocardial infarction and angina pectoris. BMC Med Genomics. 2013 May 4;6:16. doi: 10.1186/1755-8794-6-16. PMID 23641832
- [Background] Nagalla S, Shaw C, Kong X, Kondkar AA, Edelstein LC, Ma L, Chen J, McKnight GS, Lopez JA, Yang L, Jin Y, Bray MS, Leal SM, Dong JF, Bray PF. Platelet microRNA-mRNA coexpression profiles correlate with platelet reactivity. Blood. 2011 May 12;117(19):5189-97. doi: 10.1182/blood-2010-09-299719. Epub 2011 Mar 17. PMID 21415270
- [Background] Katz MG, Fargnoli AS, Williams RD, Kendle AP, Steuerwald NM, Bridges CR. MiRNAs as potential molecular targets in heart failure. Future Cardiol. 2014 Nov;10(6):789-800. doi: 10.2217/fca.14.64. PMID 25495820
- [Background] Song MA, Paradis AN, Gay MS, Shin J, Zhang L. Differential expression of microRNAs in ischemic heart disease. Drug Discov Today. 2015 Feb;20(2):223-35. doi: 10.1016/j.drudis.2014.10.004. Epub 2014 Oct 23. PMID 25461956
- [Background] Mitchell PS, Parkin RK, Kroh EM, Fritz BR, Wyman SK, Pogosova-Agadjanyan EL, Peterson A, Noteboom J, O'Briant KC, Allen A, Lin DW, Urban N, Drescher CW, Knudsen BS, Stirewalt DL, Gentleman R, Vessella RL, Nelson PS, Martin DB, Tewari M. Circulating microRNAs as stable blood-based markers for cancer detection. Proc Natl Acad Sci U S A. 2008 Jul 29;105(30):10513-8. doi: 10.1073/pnas.0804549105. Epub 2008 Jul 28. PMID 18663219